CLINICAL TRIAL: NCT01865019
Title: Pressure Controlled Versus Volume Controlled Mechanical Ventilation During Anesthesia for Living Donor Liver Transplantation Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Yassen, PROFESSOR, Mansoura University
Other Study IDs: 1981; 2013 (Other: GASTROENTEROLOGY CENTER LIVER TRANSPLANTATION ANESTHESIA TEAM)
Record Dates: First submitted 2013-04-23; First posted 2013-05-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Living Donor Liver Transplantation Recipients
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- volume controlled: volume ontrolled ventilation
  Interventions: Device: mechanical ventilation
- pressure controlled: pressure controlled ventilation
  Interventions: Device: mechanical ventilation

INTERVENTIONS:
Device: mechanical ventilation

SUMMARY:
pressure controlled ventilation will improve oxygenation indices , hemodynamics during anesthesia for living donor liver transplantation recipients ,improving postoperative graft function and decreasing postoperative pulmonary complications

ELIGIBILITY:
Inclusion Criteria:

* all living donor liver transplantation recipients scheduled

Exclusion Criteria:

* Moderate to severe restrictive pulmonary functions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: living donor liver transplantation recipients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
oxygen tension | during intraoperative period

SECONDARY OUTCOMES:
decreased postoperative pulmonary complications | one week postoperative

OTHER OUTCOMES:
improved intraoperative hemodynamics | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology center, Al Mansurah, Dakahlia Governorate, Egypt